CLINICAL TRIAL: NCT07220031
Title: Effect of Activated Charcoal on Serum Osmolality, Osmolal Gap, and Enzymatic Ethylene Glycol Assay
Status: Not yet recruiting | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2251702-2
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Osmolality Disturbance; Lab Interference
Keywords: activated charcoal; serum osmolality; osmolal gap; ethylene glycol; glycerol dehydrogenase
MeSH Terms: conditions — Anthrax | interventions — Charcoal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Charcoal: Healthy volunteers to consume activated charcoal
  Interventions: Drug: Activated Charcoal

INTERVENTIONS:
Drug: Activated Charcoal — This is the only intervention

SUMMARY:
The goal of this observational study is to determine whether a clinically relevant dose of activated charcoal raises the serum osmolality and osmolal gap in a population of healthy volunteers. Secondarily to determine whether the same dose creates a false positive result using an enzymatic assay.

1. Does a clinically relevant dose of commercially available activated charcoal raise the osmolal gap above the baseline of a healthy volunteer?
2. Does the same dose of charcoal cause a false positive enzymatic assay for ethylene glycol?

Participants will be asked to consume a dose of activated charcoal and have serial blood draws for laboratory measurements.

DETAILED DESCRIPTION:
Healthy volunteers will be recruited and informed consent obtained. Exclusion criteria include acute illness or chronic condition requiring medication which would not be appropriate to discontinue due to risk for adsorption by activated charcoal.

Participants will fast prior to the study period and will have baseline laboratory measures (BMP, osmolality, ethanol, ethylene glycol). They will drink a dose of 1g/kg (max 100g) of activated charcoal suspension (Actidose Aqua) in water. Serial laboratory measurements will be made at 0.5, 1, 2,4, and 6 hours (including osmolality, osmolal gap, and ethylene glycol measured by enzymatic assay). These values will be compared to the pre-treatment values to determine if there is a change in the osmolal gap or ethylene glycol result from baseline.

This study is funded by the SUNY Upstate Department of Emergency Medicine and is approved by the IRB of the same institution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Any medical comorbidities
* Recent illness
* Pregnancy
* Prisoners
* Non-English speaking
* Weight > 100 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Osmol Gap Change | 6 hours
  Delta serum osmolality and osmolal gap at time points 0.5, 1, 2, 4, and 6 hours after Activated charcoal given

SECONDARY OUTCOMES:
Ethylene Glycol | 6 hours
  Numeric result of ethylene glycol testing (measured by glycerol dehydrogenase assay) before and after charcoal.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Calleo, MD, Principal Investigator — Upstate Medical University
Locations (1):
- Upstate Medical University Clinical Research Unit, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robson AF, Lawson AJ, Lewis L, Jones A, George S. Validation of a rapid, automated method for the measurement of ethylene glycol in human plasma. Ann Clin Biochem. 2017 Jul;54(4):481-489. doi: 10.1177/0004563216667752. Epub 2016 Aug 17. PMID 27538769
- [Background] Rooney SL, Ehlers A, Morris C, Drees D, Davis SR, Kulhavy J, Krasowski MD. Use of a Rapid Ethylene Glycol Assay: a 4-Year Retrospective Study at an Academic Medical Center. J Med Toxicol. 2016 Jun;12(2):172-9. doi: 10.1007/s13181-015-0516-6. PMID 26553280
- [Background] Huntbach W, Moss M. Rapid availability of ethylene glycol test results with enzymatic assay. Clin Toxicol (Phila). 2024 Aug;62(8):536-538. doi: 10.1080/15563650.2024.2377281. Epub 2024 Jul 15. PMID 39007755
- [Background] Coulson L, Surla A, Tran V, Hoggett K. Severe glycerol intoxication mimicking toxic alcohol ingestion following large volume consumption of vanilla essence. Clin Toxicol (Phila). 2022 Nov;60(11):1248-1250. doi: 10.1080/15563650.2022.2114911. Epub 2022 Aug 31. PMID 36043532
- [Background] Burkitt JM, Haskins SC, Aldrich J, Jandrey KE, Rezende ML, Boyle JE. Effects of oral administration of a commercial activated charcoal suspension on serum osmolality and lactate concentration in the dog. J Vet Intern Med. 2005 Sep-Oct;19(5):683-6. doi: 10.1892/0891-6640(2005)19[683:eooaoa]2.0.co;2. PMID 16231712